CLINICAL TRIAL: NCT03908528
Title: Role of Alpha-Lipoic Acid Against Chemotherapy Induced Toxicities in Breast Cancer Patients
Brief Title: Alpha-Lipoic Acid in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Principal Investigator, Rehab Werida, Lecturer, Damanhour University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Alpha-Lipoic Acid
Record Dates: First submitted 2019-03-29; First posted 2019-04-09 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer; Chemotherapeutic Toxicity
Keywords: alpha-lipoic acid; taxol; Adriamycin; cyclophosphamide; breast cancer; Brain Natriuretic Peptide (BNP).; Neurotensin; TNF-alpha
MeSH Terms: conditions — Breast Neoplasms | interventions — Thioctic Acid; Drug Therapy; Doxorubicin

STUDY DESIGN:
Intervention Model Description: Double-blind study, Patients will be classified as follow:
  * Group one: 32 patients will receive four cycles of AC followed by weekly taxol for 12 weeks plus placebo.
  * Group two: 32 patients will receive four cycles of AC followed by weekly taxol for 12 weeks plus oral 600 mg alpha lipoic acid (ALA) once daily.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy plus Placebo for six Months (Experimental): • Group one: 32 patients will receive four cycles of AC followed by weekly taxol for 12 weeks plus Placebo.
  Interventions: Other: Placebo Plus Chemotherapy (doxorubicin (also known as Adriamycin) plus cyclophosphamide followed by taxol)
- Chemotherapy plus alpha lipoic acid for six Months (Experimental): • Group two: 32 patients will receive four cycles of AC followed by weekly taxol for 12 weeks in addition to oral 600 mg alpha lipoic acid (ALA) once daily.
  Interventions: Dietary Supplement: Alpha-lipoic acid Plus Chemotherapy (doxorubicin (also known as Adriamycin) plus cyclophosphamide followed by taxol)

INTERVENTIONS:
Dietary Supplement: Alpha-lipoic acid Plus Chemotherapy (doxorubicin (also known as Adriamycin) plus cyclophosphamide followed by taxol) — 600 mg Alpha-lipoic acid daily (an antioxidant that's in many foods, and it's made naturally in the investigator's bodies) with four cycles of doxorubicin (also known as Adriamycin) plus cyclophosphamide followed by weekly taxol for 12 weeks..
  Other Names: Thiotacid 600 mg
  Arms: Chemotherapy plus alpha lipoic acid for six Months
Other: Placebo Plus Chemotherapy (doxorubicin (also known as Adriamycin) plus cyclophosphamide followed by taxol) — Placebo with four cycles of doxorubicin (also known as Adriamycin) plus cyclophosphamide followed by weekly taxol for 12 weeks.
  Other Names: placebo
  Arms: Chemotherapy plus Placebo for six Months

SUMMARY:
• Investigate the ability of alpha lipoic acid to counter act anthracycline associated cardiotoxicity and cumulative taxens-related PN in patients with breast cancer.

DETAILED DESCRIPTION:
Fifty breast cancer patients with stage from stage I to stage III will be involved in this study. Staging is done according to the American joint committee on cancer: TNM staging of breast cancer.

* All participants will be recruited from Tanta Oncology Center. The study will be approved by Research Ethics Committee of Damanhour University. All participants will give their consent.
* All 64 patients will be scheduled to receive 4 cycles of AC: cycled every 21 days followed by weekly cycle of taxol for 12 weeks.

Patients will be classified as follow:

* Group one: 32 patients will receive four cycles of AC followed by weekly taxol for 12 weeks plus placebo.
* Group two: 32 patients will receive the same regimen as group 1 in addition to oral 600 mg alpha lipoic acid (ALA) once daily.

All patients will be submitted to:

1. Full patient history and clinical examination.
2. Venous blood will be collected before the first cycle of chemotherapy and after the last cycle of chemotherapy.

1- Cardio-toxcity assessment: i. Echo-cardiogram. ii. Troponin I. iii. The Brain Natriuretic Peptide (BNP). 2- Neurotoxicity assessment: i. National Cancer Institute common Terminology criteria for Adverse Effect grading: NCI-CTCAE version 4.0.

ii. Neurotoxicity questionnaire from the validated Functional Assessment of cancer therapy/gynecologic oncology group taxane specific neurotoxicity questionnaire: FACT-Taxane.

iii. Neurotensin 3- Oxidative stress and inflammatory markers: i. Malondialdehyde (MDA). ii. TNF-alpha

ELIGIBILITY:
Inclusion Criteria:

1. All patients age ≥ 18 and < 70 years old with confirmed stage from stage I to stage III.
2. No evidence of metastases at initial assessment.
3. Patients has to have a good performance status (ECOG 0-2) according to Eastern Cooperative Oncology Group (ECOG) score.
4. Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin level ≥ 10g/dL).
5. Patients with adequate liver function (serum creatinine < 1.5 mg/dL) and adequate renal function (serum creatinine < 1.5 mg/dL, creatinine clearance (CrCl) > 45 ml/min).
6. Either pre operative or post operative chemotherapy are allowed.

Exclusion Criteria:

1. Evidence of metastases at initial assessment.
2. Pregnancy or breast-feeding patients.
3. Prior exposure to neurotoxic chemotherapy was not allowed (no carboplatin, vincristine, vinblastine, paclitaxel, or docetaxol ) for 6 months prior study treatment.
4. Clinical evidence of serious cardiac illness (myocardial dysfunctional, angina pectoris requiring anti-angina medication, poorly controlled hypertension, and uncontrolled arrhythmias).
5. Patients with a reduced cardiac output with a left ventricular ejection fraction (LVEF) ejection fraction < 50%.
6. Patients who had evidence of pre-existing peripheral neuropathy resulting from another reason (diabetes).
7. Patients with a history of allergy to alpha-lipoic acid.
8. Concomitant use of multivitamins (vitamin E), opioids, anticonvulsants, tricyclic antidepressants, other neuropathic pain medication modifying agents (e.g., gabapentin, lamotrigine, carbamazepine, phenytoin, or tricyclic antidepressants) are not allowed

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Cardiotoxcity assessment | six months
  serum Brain Natriuretic Peptide (BNP) level
Neurotoxicity assessment | six months
  Neurotensin level
oxidative stress and inflammatory markers | six months
  TNF-alpha level
MDA | six months
  Malondialdehyde

CONTACTS AND LOCATIONS:
Overall Officials: Reham A Elshafiey, PharmD, Principal Investigator — Damanhour University
Locations (1):
- Tanta Oncology Center, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapoor S. The Anti-neoplastic Effects of Alpha-Lipoic Acid: Clinical Benefits in System Tumors besides Lung Carcinomas. Korean J Thorac Cardiovasc Surg. 2013 Apr;46(2):162-3. doi: 10.5090/kjtcs.2013.46.2.162. Epub 2013 Apr 9. No abstract available. PMID 23614108
- [Derived] Werida RH, Elshafiey RA, Ghoneim A, Elzawawy S, Mostafa TM. Role of alpha-lipoic acid in counteracting paclitaxel- and doxorubicin-induced toxicities: a randomized controlled trial in breast cancer patients. Support Care Cancer. 2022 Sep;30(9):7281-7292. doi: 10.1007/s00520-022-07124-0. Epub 2022 May 21. PMID 35596774